CLINICAL TRIAL: NCT00893035
Title: Multicenter Prospective Evaluation of a Predictive Test of Late Toxicities After Radiotherapy by the Rate of Radiation Induced CD8 T-Lymphocyte Apoptosis: Application to Breast and Prostate Cancers.
Brief Title: Evaluation of an Apoptotic Test for Predicting Late Toxicities After Radiotherapy in Breast and Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC 2005 DA
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Radiotherapy; Late side effects; Predictive assay
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intermediate prognosis prostate cancer: Intermediate prognosis prostate cancer
- Breast cancer: conservative treatment and age<60 Boost irradiation and age>60

SUMMARY:
The primary objective of this study is to evaluate the prediction of late toxicity by the radiation induced CD8 T-lymphocyte apoptosis

DETAILED DESCRIPTION:
The two cancer sites concerned by this trial are intermediate risk prostate cancer treated with conformational radiotherapy with or without intensity modulation, and breast cancer patients treated with adjuvant radiotherapy after breast conservative surgery for patients aged under 60 years of age. The identification of 5% of patients at risk of severe toxicity should allow to deliver high dose radiotherapy among 95% of patients with a lower risk of severe late complications.

ELIGIBILITY:
Inclusion Criteria for prostate cancer patients:

* localised prostate cancer, histologically proven
* Absence of metastases (M0) : normal bone scintigraphy
* Absence of radiological lymph node invasion (N0).
* Clinical Stage : T ≥ T1c-T2a and < T3b Or T1b or c with PSA ≤ 10 ng/ml . Or T1b or c with Gleason ≥ 6
* PSA < 30 ng/ml.
* Signs and symptoms according to NCI/CTC v3.0 < grade 2
* ECOG Performance status ≤ 1
* Absence of hip prothesis
* Absence de endopenian stent
* Patient aged > 18 and < 80
* Patient affiliated with social security
* Written informed consent, dated and signed

Exclusion Criteria for prostate cancer patients:

* Antecedents of invasive cancer (unless if treated more than 5 years ago without evolution) except basocellular carcinoma
* positive biopsy of seminal vesicle
* PSA ≥ 30 ng/ml for two successive dosages
* Previous pelvic irradiation
* Previous radical prostatectomy for cancer
* Patients with another systemic disease (cardiovascular, renal, hepatic, pulmonary embolism, etc.) non stabilised or generalised sclerodermitis.
* Patients known to be HIV seropositive (no specific test is necessary for defining eligibility)
* Known homozygote ATM (Ataxy telangiectasy) mutation
* Impossibility for a correct follow up (for social family or geographical reasons)
* Patients incapable of providing consent, protected majors, vulnerable persons
* Patients participating in other clinical trials

Inclusion Criteria for breast cancer patients:

* Breast Conservative surgery
* Non metastatic, M0
* negative surgical margins
* T1, T2; negative sentinel lymph node N0, N1 or N2.
* Signs and symptoms according to NCI/CTC v3.0 < grade 2
* Patient aged over 18 years and less than 60 or more than 60 with an indication for boost irradiation.
* Patient affiliated with social security
* Written informed consent, dated and signed

Exclusion Criteria for breast cancer patients:

* Metastatic patients
* Bilateral breast cancer (concomitant or previous) except in situ
* T4 or N3 or treated by mastectomy
* Patients with chemotherapy or neoadjuvant hormonotherapy
* Patients with a previous other cancer within the last 5 years EXCEPT basocellular carcinoma of the skin or in situ cancer of the uterus.
* Patients with another systemic disease (cardiovascular, renal, hepatic, pulmonary embolism, etc.) non stabilised or generalised sclerodermia.
* Pregnant or breast feeding women
* Patients known to be HIV seropositive (no specific test is necessary for defining eligibility)
* Known homozygote ATM (Ataxy telangiectasy) mutation
* Impossibility for a correct follow up (for social family or geographical reasons)
* Patients incapable of providing consent, protected majors, vulnerable persons
* Patients participating in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated in a cancer center
Sampling Method: Non-Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2006-06; Primary Completion 2015-12 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Late complications | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Azria, Principal Investigator — CRLC Val d'Aurelle
Locations (1):
- CRLC Val d'Aurelle, Montpellier, France

REFERENCES:
- [Background] Arriagada R, Mouriesse H, Sarrazin D, Clark RM, Deboer G. Radiotherapy alone in breast cancer. I. Analysis of tumor parameters, tumor dose and local control: the experience of the Gustave-Roussy Institute and the Princess Margaret Hospital. Int J Radiat Oncol Biol Phys. 1985 Oct;11(10):1751-7. doi: 10.1016/0360-3016(85)90027-6. PMID 4044337
- [Background] Azria D, Gourgou S, Sozzi WJ, Zouhair A, Mirimanoff RO, Kramar A, Lemanski C, Dubois JB, Romieu G, Pelegrin A, Ozsahin M. Concomitant use of tamoxifen with radiotherapy enhances subcutaneous breast fibrosis in hypersensitive patients. Br J Cancer. 2004 Oct 4;91(7):1251-60. doi: 10.1038/sj.bjc.6602146. PMID 15328527
- [Background] Bartelink H, Horiot JC, Poortmans P, Struikmans H, Van den Bogaert W, Barillot I, Fourquet A, Borger J, Jager J, Hoogenraad W, Collette L, Pierart M; European Organization for Research and Treatment of Cancer Radiotherapy and Breast Cancer Groups. Recurrence rates after treatment of breast cancer with standard radiotherapy with or without additional radiation. N Engl J Med. 2001 Nov 8;345(19):1378-87. doi: 10.1056/NEJMoa010874. PMID 11794170
- [Background] Buchholz TA. Finding our sensitive patients. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):547-8. doi: 10.1016/s0360-3016(99)00255-2. No abstract available. PMID 10524402
- [Background] Cesaretti JA, Stock RG, Lehrer S, Atencio DA, Bernstein JL, Stone NN, Wallenstein S, Green S, Loeb K, Kollmeier M, Smith M, Rosenstein BS. ATM sequence variants are predictive of adverse radiotherapy response among patients treated for prostate cancer. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):196-202. doi: 10.1016/j.ijrobp.2004.09.031. PMID 15629612
- [Background] Crompton NE, Ozsahin M. A versatile and rapid assay of radiosensitivity of peripheral blood leukocytes based on DNA and surface-marker assessment of cytotoxicity. Radiat Res. 1997 Jan;147(1):55-60. PMID 8989370
- [Background] Crompton NE, Shi YQ, Emery GC, Wisser L, Blattmann H, Maier A, Li L, Schindler D, Ozsahin H, Ozsahin M. Sources of variation in patient response to radiation treatment. Int J Radiat Oncol Biol Phys. 2001 Feb 1;49(2):547-54. doi: 10.1016/s0360-3016(00)01477-2. PMID 11173153
- [Background] Delanian S, Balla-Mekias S, Lefaix JL. Striking regression of chronic radiotherapy damage in a clinical trial of combined pentoxifylline and tocopherol. J Clin Oncol. 1999 Oct;17(10):3283-90. doi: 10.1200/JCO.1999.17.10.3283. PMID 10506631
- [Background] Delanian S, Porcher R, Balla-Mekias S, Lefaix JL. Randomized, placebo-controlled trial of combined pentoxifylline and tocopherol for regression of superficial radiation-induced fibrosis. J Clin Oncol. 2003 Jul 1;21(13):2545-50. doi: 10.1200/JCO.2003.06.064. PMID 12829674
- [Background] Denis F, Garaud P, Bardet E, Alfonsi M, Sire C, Germain T, Bergerot P, Rhein B, Tortochaux J, Oudinot P, Calais G. Late toxicity results of the GORTEC 94-01 randomized trial comparing radiotherapy with concomitant radiochemotherapy for advanced-stage oropharynx carcinoma: comparison of LENT/SOMA, RTOG/EORTC, and NCI-CTC scoring systems. Int J Radiat Oncol Biol Phys. 2003 Jan 1;55(1):93-8. doi: 10.1016/s0360-3016(02)03819-1. PMID 12504040
- [Background] Dewey WC, Ling CC, Meyn RE. Radiation-induced apoptosis: relevance to radiotherapy. Int J Radiat Oncol Biol Phys. 1995 Nov 1;33(4):781-96. doi: 10.1016/0360-3016(95)00214-8. PMID 7591884
- [Background] Dubray B. [Late complications of radiotherapy. Role of the time factor]. Bull Cancer Radiother. 1995;82(2):98-100. No abstract available. French. PMID 7546901
- [Background] Emami B, Lyman J, Brown A, Coia L, Goitein M, Munzenrider JE, Shank B, Solin LJ, Wesson M. Tolerance of normal tissue to therapeutic irradiation. Int J Radiat Oncol Biol Phys. 1991 May 15;21(1):109-22. doi: 10.1016/0360-3016(91)90171-y. PMID 2032882
- [Background] Fine JP. Regression modeling of competing crude failure probabilities. Biostatistics. 2001 Mar;2(1):85-97. doi: 10.1093/biostatistics/2.1.85. PMID 12933558
- [Background] Floyd DN, Cassoni AM. Intrinsic radiosensitivity of adult and cord blood lymphocytes as determined by the micronucleus assay. Eur J Cancer. 1994;30A(5):615-20. doi: 10.1016/0959-8049(94)90531-2. PMID 8080675
- [Background] Hoeller U, Borgmann K, Bonacker M, Kuhlmey A, Bajrovic A, Jung H, Alberti W, Dikomey E. Individual radiosensitivity measured with lymphocytes may be used to predict the risk of fibrosis after radiotherapy for breast cancer. Radiother Oncol. 2003 Nov;69(2):137-44. doi: 10.1016/j.radonc.2003.10.001. PMID 14643950
- [Background] Hsieh FY, Lavori PW. Sample-size calculations for the Cox proportional hazards regression model with nonbinary covariates. Control Clin Trials. 2000 Dec;21(6):552-60. doi: 10.1016/s0197-2456(00)00104-5. PMID 11146149
- [Background] Iannuzzi CM, Atencio DP, Green S, Stock RG, Rosenstein BS. ATM mutations in female breast cancer patients predict for an increase in radiation-induced late effects. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):606-13. doi: 10.1016/s0360-3016(01)02684-0. PMID 11849780
- [Background] Jacob R, Hanlon AL, Horwitz EM, Movsas B, Uzzo RG, Pollack A. Role of prostate dose escalation in patients with greater than 15% risk of pelvic lymph node involvement. Int J Radiat Oncol Biol Phys. 2005 Mar 1;61(3):695-701. doi: 10.1016/j.ijrobp.2004.06.023. PMID 15708247
- [Background] Johansen J, Bentzen SM, Overgaard J, Overgaard M. Relationship between the in vitro radiosensitivity of skin fibroblasts and the expression of subcutaneous fibrosis, telangiectasia, and skin erythema after radiotherapy. Radiother Oncol. 1996 Aug;40(2):101-9. doi: 10.1016/0167-8140(96)01777-x. PMID 8884963
- [Background] Kiltie AE, Ryan AJ, Swindell R, Barber JB, West CM, Magee B, Hendry JH. A correlation between residual radiation-induced DNA double-strand breaks in cultured fibroblasts and late radiotherapy reactions in breast cancer patients. Radiother Oncol. 1999 Apr;51(1):55-65. doi: 10.1016/s0167-8140(99)00030-4. PMID 10386717
- [Background] Lartigau E, Dubray B, Mornex F. [Biological mechanisms of late effects of ionizing radiations]. Cancer Radiother. 1997;1(6):669-76. doi: 10.1016/s1278-3218(97)82943-5. French. PMID 9614881
- [Background] Latouche A, Porcher R, Chevret S. Sample size formula for proportional hazards modelling of competing risks. Stat Med. 2004 Nov 15;23(21):3263-74. doi: 10.1002/sim.1915. PMID 15490425
- [Background] Ozsahin M, Ozsahin H, Shi Y, Larsson B, Wurgler FE, Crompton NE. Rapid assay of intrinsic radiosensitivity based on apoptosis in human CD4 and CD8 T-lymphocytes. Int J Radiat Oncol Biol Phys. 1997 May 1;38(2):429-40. doi: 10.1016/s0360-3016(97)00038-2. PMID 9226332
- [Background] Pepe MS, Mori M. Kaplan-Meier, marginal or conditional probability curves in summarizing competing risks failure time data? Stat Med. 1993 Apr 30;12(8):737-51. doi: 10.1002/sim.4780120803. PMID 8516591
- [Background] Pollack A, Smith LG, von Eschenbach AC. External beam radiotherapy dose response characteristics of 1127 men with prostate cancer treated in the PSA era. Int J Radiat Oncol Biol Phys. 2000 Sep 1;48(2):507-12. doi: 10.1016/s0360-3016(00)00620-9. PMID 10974469
- [Background] Pollack A, Zagars GK, Smith LG, Lee JJ, von Eschenbach AC, Antolak JA, Starkschall G, Rosen I. Preliminary results of a randomized radiotherapy dose-escalation study comparing 70 Gy with 78 Gy for prostate cancer. J Clin Oncol. 2000 Dec 1;18(23):3904-11. doi: 10.1200/JCO.2000.18.23.3904. PMID 11099319
- [Background] Radford IR, Murphy TK. Radiation response of mouse lymphoid and myeloid cell lines. Part III. Different signals can lead to apoptosis and may influence sensitivity to killing by DNA double-strand breakage. Int J Radiat Biol. 1994 Feb;65(2):229-39. doi: 10.1080/09553009414550261. PMID 7907120
- [Background] Romestaing P, Lehingue Y, Carrie C, Coquard R, Montbarbon X, Ardiet JM, Mamelle N, Gerard JP. Role of a 10-Gy boost in the conservative treatment of early breast cancer: results of a randomized clinical trial in Lyon, France. J Clin Oncol. 1997 Mar;15(3):963-8. doi: 10.1200/JCO.1997.15.3.963. PMID 9060534
- [Background] Slonina D, Gasinska A. Intrinsic radiosensitivity of healthy donors and cancer patients as determined by the lymphocyte micronucleus assay. Int J Radiat Biol. 1997 Dec;72(6):693-701. doi: 10.1080/095530097142852. PMID 9416792
- [Background] Stone HB, Coleman CN, Anscher MS, McBride WH. Effects of radiation on normal tissue: consequences and mechanisms. Lancet Oncol. 2003 Sep;4(9):529-36. doi: 10.1016/s1470-2045(03)01191-4. PMID 12965273
- [Background] Thames HD, Hendry JH, Moore JV, Ang KK, Travis EL. The high steepness of dose-response curves for late-responding normal tissues. Radiother Oncol. 1989 May;15(1):49-53. doi: 10.1016/0167-8140(89)90117-5. PMID 2748942
- [Background] Trotti A, Byhardt R, Stetz J, Gwede C, Corn B, Fu K, Gunderson L, McCormick B, Morrisintegral M, Rich T, Shipley W, Curran W. Common toxicity criteria: version 2.0. an improved reference for grading the acute effects of cancer treatment: impact on radiotherapy. Int J Radiat Oncol Biol Phys. 2000 Apr 1;47(1):13-47. doi: 10.1016/s0360-3016(99)00559-3. PMID 10758303
- [Background] Trotti A, Colevas AD, Setser A, Rusch V, Jaques D, Budach V, Langer C, Murphy B, Cumberlin R, Coleman CN, Rubin P. CTCAE v3.0: development of a comprehensive grading system for the adverse effects of cancer treatment. Semin Radiat Oncol. 2003 Jul;13(3):176-81. doi: 10.1016/S1053-4296(03)00031-6. PMID 12903007
- [Background] TROWELL OA. The sensitivity of lymphocytes to ionising radiation. J Pathol Bacteriol. 1952 Oct;64(4):687-704. doi: 10.1002/path.1700640403. No abstract available. PMID 13000583
- [Background] Withers HR, Taylor JM, Maciejewski B. Treatment volume and tissue tolerance. Int J Radiat Oncol Biol Phys. 1988 Apr;14(4):751-9. doi: 10.1016/0360-3016(88)90098-3. PMID 3350731
- [Background] Zelefsky MJ, Fuks Z, Hunt M, Yamada Y, Marion C, Ling CC, Amols H, Venkatraman ES, Leibel SA. High-dose intensity modulated radiation therapy for prostate cancer: early toxicity and biochemical outcome in 772 patients. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1111-6. doi: 10.1016/s0360-3016(02)02857-2. PMID 12128109
- [Result] Lacombe J, Brengues M, Mange A, Bourgier C, Gourgou S, Pelegrin A, Ozsahin M, Solassol J, Azria D. Quantitative proteomic analysis reveals AK2 as potential biomarker for late normal tissue radiotoxicity. Radiat Oncol. 2019 Aug 9;14(1):142. doi: 10.1186/s13014-019-1351-8. PMID 31399108
- [Result] Azria D, Riou O, Castan F, Nguyen TD, Peignaux K, Lemanski C, Lagrange JL, Kirova Y, Lartigau E, Belkacemi Y, Bourgier C, Rivera S, Noel G, Clippe S, Mornex F, Hennequin C, Kramar A, Gourgou S, Pelegrin A, Fenoglietto P, Ozsahin EM. Radiation-induced CD8 T-lymphocyte Apoptosis as a Predictor of Breast Fibrosis After Radiotherapy: Results of the Prospective Multicenter French Trial. EBioMedicine. 2015 Oct 25;2(12):1965-73. doi: 10.1016/j.ebiom.2015.10.024. eCollection 2015 Dec. PMID 26844275
- [Result] Bourgier C, Castan F, Riou O, Nguyen TD, Peignaux K, Lemanski C, Lagrange JL, Kirova Y, Lartigau E, Belkacemi Y, Rivera S, Noel G, Clippe S, Mornex F, Hennequin C, Gourgou S, Brengues M, Fenoglietto P, Ozsahin EM, Azria D. Impact of adjuvant hormonotherapy on radiation-induced breast fibrosis according to the individual radiosensitivity: results of a multicenter prospective French trial. Oncotarget. 2018 Mar 2;9(21):15757-15765. doi: 10.18632/oncotarget.24606. eCollection 2018 Mar 20. PMID 29644007
- [Result] Touraine C, Winter A, Castan F, Azria D, Gourgou S. Time-Dependent ROC Curve Analysis for Assessing the Capability of Radiation-Induced CD8 T-Lymphocyte Apoptosis to Predict Late Toxicities after Adjuvant Radiotherapy of Breast Cancer Patients. Cancers (Basel). 2023 Sep 22;15(19):4676. doi: 10.3390/cancers15194676. PMID 37835370